CLINICAL TRIAL: NCT04070612
Title: National Prospective Cohort for Monitoring Children With Severe Autoimmune Cytopenia
Acronym: BIOCEREVANCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2005/18
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cytopenia; Autoimmune Haemolytic Anaemia; Thrombocytopenic Purpura, Immune
Keywords: Children
MeSH Terms: conditions — Cytopenia; Anemia, Hemolytic, Autoimmune; Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children with autoimmune haemolytic anemia: A blood sample of 2 times 2 to 5 ml additional maximum
  Interventions: Other: Blood sample
- Children with Evans syndrome: A blood sample of 2 times 2 to 5 ml additional maximum
  Interventions: Other: Blood sample
- Children with Immune thrombocytopenic purpura: A blood sample of 2 times 2 to 5 ml additional maximum
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample of 2 times 2 to 5 ml additional maximum

SUMMARY:
This study aims to study prospectively the clinical and paraclinical evolution and prognostic factors of autoimmune haemolytic anemias, Evans syndromes and chronic immunological thrombocytopenic purpura of children in France.

DETAILED DESCRIPTION:
These autoimmune haematological diseases are rare diseases affecting the child, often very young, and serious and potentially life-threatening. International literature data are scarce, and include individual cases or small series.

They do not allow to determine an optimal therapeutic strategy in case of escape from the first-line treatments. Existing treatments (long-term corticosteroid therapy, immunoglobulins, splenectomy, immunosuppressants, chemotherapies, and more recently anti-CD20 antibodies) are inconsistently effective, and often associated with serious side effects.

The seriousness of these diseases, the therapeutic difficulties, and the absence of a targeted research project in France, led to the implementation of this study.

This study aims to study prospectively the clinical and paraclinical evolution and prognostic factors of autoimmune haemolytic anemias, Evans syndromes and chronic immunological thrombocytopenic purpura of children in France.

ELIGIBILITY:
Inclusion Criteria:

* Age strictly below 18 years of age at initial diagnosis
* Affiliate child or beneficiary of a social security scheme
* Child residing in metropolitan France
* Diagnosis of autoimmune haemolytic anemias, Evans syndrome and / or chronic Immune thrombocytopenic purpura
* Free, informed, written and signed consent

Exclusion Criteria:

* Diagnosis of constitutional haemolytic anemia
* Diagnosis of platelet constitutional disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2007-04-04 (Actual); Primary Completion 2012-06-08 (Actual); Study Completion 2012-06-08 (Actual)

PRIMARY OUTCOMES:
Complete sustainable remission (yes/no) for children with autoimmune haemolytic anemias | At the screening
  Absence of clinical signs of anemia (grade 0) And Hemoglobin > 11 g / dl And reticulocytes <120,000 / mm3 And haptoglobin> 10 mg / dl And bilirubin <10 mg / l or 17 μmol / l And no specific treatment for at least 12 months
complete remission (yes/no) for children with autoimmune haemolytic anemias | At the screening
  Absence of clinical signs of anemia (grade 0) And Hemoglobin> 11 g / dl And reticulocytes <120,000 / mm3 Regardless of the level of haptoglobin or bilirubin And specific treatment in progress or interrupted for less than 12 months
partial remission (yes/no) for children with autoimmune haemolytic anemias | At the screening
  Clinical Signs of Anemia (Grade 1 or 2) Or Hemoglobin from 7 to 11 g / dl Or reticulocytes> 120,000 / mm3 Regardless of the level of haptoglobin or bilirubin
no response (yes/no) for children with autoimmune haemolytic anemias | At the screening
  Clinical Signs of Severe Anemia (Grade 3 or More) Or Hemoglobin <7 g / dl
deceased patient (yes/no) for children with autoimmune haemolytic anemias | At the screening
  Death yes/no
Complete sustainable remission (yes/no) for children with chronic immunologic thrombocytopenic purpura | At the screening
  Absence of clinical signs of haemorrhage (grade 0) And platelets> 100,000 / mm3 And no specific treatment for at least 12 months
complete remission (yes/no) for children with chronic immunologic thrombocytopenic purpura | At the screening
  Absence of clinical signs of haemorrhage (grade 0) And platelets> 100,000 / mm3 And specific treatment in progress or interrupted for less than 12 months
partial remission (yes/no) for children with chronic immunologic thrombocytopenic purpura | At the screening
  Clinical Signs of Hemorrhage (Grade 1 or 2) Or platelets between 30,000 and 100,000 / mm3
no response (yes/no) for children with chronic immunologic thrombocytopenic purpura | At the screening
  Clinical Signs of Severe Hemorrhage (Grade 3 or Greater) Or Platelets <30,000 / mm3
deceased patient (yes/no) for children with chronic immunologic thrombocytopenic purpura | At the screening
  Death yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Yves PEREL, Pr, Principal Investigator — Bordeaux University Hsopital

IPD SHARING:
Plan to Share IPD: No